CLINICAL TRIAL: NCT06825689
Title: Unidos Contra el VPH: Screening Preference and Uptake of HPV Self-sampling Among Latinxs Along the US-Mexico Border
Brief Title: Unidos Contra el VPH
Acronym: Unidos
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Jessica Calderon-Mora, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CPRIT-RP240208; STUDY00005986 (Other: University of Texas at Austin Dell Medical School)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Human Papilloma Virus (HPV); Cervical Cancers
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Group 1: Urine Self-Sampling (Experimental): Participants in this group receive a kit with a urine sample cup to use at home, instructions explaining how to take the sample and a pre-paid mailing box to mail the urine sample to the lab.
  Interventions: Device: Self-sampling with urine
- Group 2: Swab Self-Sampling (Experimental): Participants in this group receive a kit with a vaginal swab and collection tube to use at home, instructions explaining how to take the sample and a pre-paid mailing box to mail the sample to the lab.
  Interventions: Device: Self-sampling with swab
- Group 3: In-Clinic Co-Testing (Active Comparator): Participants in this group are scheduled for an in-clinic Pap smear/HPV co-testing appointment.
  Interventions: Device: In-clinic Pap/HPV co-testing

INTERVENTIONS:
Device: Self-sampling with urine — Urine is self-collected at home using a urine sample cup.
  Arms: Group 1: Urine Self-Sampling
Device: Self-sampling with swab — A vaginal cell sample is self-collected at home using a swab and collection tube.
  Arms: Group 2: Swab Self-Sampling
Device: In-clinic Pap/HPV co-testing — Cervico-vaginal cell samples are collected by a clinician during a Pap smear/HPV co-test appointment.
  Arms: Group 3: In-Clinic Co-Testing

SUMMARY:
The purpose of the Unidos Contra el VPH study is to help find options to screen, or check, for cervical cancer that individuals can do at home to help prevent and detect cervical cancer early. Usually, people get screened for cervical cancer with a Pap smear and human papillomavirus (HPV) test by a health care provider. This is not always easy for individuals who are not able to get to a clinic or feel uncomfortable having the procedure done. That is why we want to find other ways that may be easier and more comfortable for people to be screened for cervical cancer.

The two main questions the study aims to answer are:

1. How do the following three cervical cancer screening methods compare for improving screening completion rates?

   o In-home HPV self-sampling with a vaginal swab
   * In-home HPV self-sampling with urine testing
   * In-clinic traditional Pap smear with HPV test
2. What are participant beliefs and preferences regarding these three screening methods?

   Participants in the study will be randomly assigned to one of three groups. This means each person has an equal chance of being placed in any group. They will also complete two surveys as part of the study. The three screening method groups are described below:

   Group 1: Urine Self-Sampling
   * Participants in this group will receive a kit with a urine sample cup to use at home, instructions explaining how to take the sample and a pre-paid mailing box to mail the urine sample to the lab.

   Group 2: Vaginal Swab Self-Sampling o Participants in this group will receive a kit with a vaginal swab and collection tube to use at home, instructions explaining how to take the sample and a pre-paid mailing box to mail the sample to the lab.

   Group 3: In-Clinic Screening
   * An in-clinic co-testing appointment is scheduled for a Pap smear and HPV test done together at Project Vida Health Center.

   By comparing these approaches, this study aims to improve access to cervical cancer screening and provide better options for those who face barriers to clinic-based screening.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a cervix who are 30-65 years and have not undergone a Pap test in at least three years.

Exclusion Criteria:

* Having had a hysterectomy or a personal history of cervical cancer.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 735 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of Completion Rates Among Three Cervical Cancer Screening Methods | Screening completion within 60 days of enrollment
  This study will compare the effectiveness of three cervical cancer screening methods in achieving screening completion. Participants will be randomized to one of the following groups:
  In-home HPV self-sampling using a urine sample In-home HPV self-sampling using a cervico-vaginal swab In-clinic cervical cancer screening via clinician-collected HPV and Pap test
  The primary outcome will be the screening completion rate-- the proportion of participants who successfully complete their assigned screening method within the study period.

SECONDARY OUTCOMES:
Comparison of Participant Beliefs and Preferences for HPV Self-Collection Versus Clinician-Collected Samples | Participants will complete surveys at two time points: baseline (at enrollment) and follow-up (within 2 weeks of screening completion).
  We will assess participant beliefs and preferences regarding three cervical cancer screening methods: (1) in-home HPV self-sampling using urine, (2) in-home HPV self-sampling using a vaginal swab, and (3) in-clinic clinician-collected samples. Participants will complete surveys measuring their perceptions, acceptability, and preferences for the different screening options. The surveys include items based on Health Belief Model constructs such as perceived susceptibility, severity, benefits, barriers, and self-efficacy. Test preference will be measured on ease, pain, embarrassment, confidence in screening method, fear of harm, and convenience.

CONTACTS AND LOCATIONS:
Locations (1):
- Project Vida Health Center, El Paso, Texas, United States